CLINICAL TRIAL: NCT00420017
Title: Prevention of Atrial Fibrillation Following Thoracoabdominal Esophagectomy Surgery
Brief Title: Prevention of Atrial Fibrillation Following Esophagectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other); Indiana University Health (Other)
Responsible Party: Principal Investigator, James E. Tisdale, Professor and Interim Head, Department of Pharmacy Practice, Purdue University, and Adjunct Professor, School of Medicine, Indiana University, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0510-23
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Results first posted 2013-02-06 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Atrial Fibrillation; Esophagectomy
Keywords: Amiodarone; Atrial fibrillation; Surgical procedures, thoracic
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amiodarone (Experimental): Intravenous amiodarone
  Interventions: Drug: Amiodarone
- Control (Other): Control
  Interventions: Other: Control

INTERVENTIONS:
Drug: Amiodarone — Intravenous amiodarone continuous infusion x 4 days
  Arms: Amiodarone
Other: Control — No amiodarone
  Arms: Control

SUMMARY:
The investigators hypothesize that the medication amiodarone decreases the incidence of atrial fibrillation (AF) following esophagectomy surgery. Their specific aims are to:

Determine the effectiveness of amiodarone for the prevention of AF following esophagectomy surgery; Determine the influence of the prevention of AF following esophagectomy surgery on post-surgical duration of stay in the Intensive Care Unit ICU)and duration of post-surgical hospital stay; and Determine the safety of amiodarone for the prevention of AF following esophagectomy surgery.

DETAILED DESCRIPTION:
Thousands of patients undergo major esophagectomy surgery in the United States each year, during which all or a portion of the esophagus is removed. A major complication of these surgeries is the occurrence of an irregular heartbeat known as atrial fibrillation (AF), which develops in up to 40% of patients undergoing these procedures. AF is characterized by rapid, irregular, chaotic beating of the two smaller chambers of the heart (the atria), leading to rapid, irregular beating of the two larger chambers (the ventricles). The average time to occurrence of post-surgical AF is 2-3 days following surgery. AF occurring following esophagectomy can result in extremely rapid heart rates, as fast as 150-200 beats per minute, and may be associated with serious consequences, including severely low blood pressure and potentially debilitating stroke. Further, the risk of death following esophagectomy is significantly higher in patients who develop AF compared with those who do not. Therefore, the occurrence of this irregular heartbeat following esophagectomy is associated with severe, potentially life-threatening consequences. Prevention of this irregular heartbeat in these patients may therefore be very important.

Amiodarone is a medication that is known to be effective for prevention and treatment of AF that occurs in patients who have not undergone surgery. In addition, amiodarone has been shown to be effective for prevention of AF following open-chest heart surgery. However, the use of medications for prevention of AF following esophagectomy has not been well studied, and amiodarone has not been studied in a controlled trial for the prevention of AF in this population. In addition, amiodarone is associated with side effects, and it is important to determine the safety of this medication when used in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Males or females over the age of 40
* Scheduled to undergo esophagectomy

Exclusion Criteria:

* History of atrial fibrillation
* Prior severe side effects from amiodarone
* Elevated liver enzymes >3 times the upper limit of normal (UNL)
* Corrected QT interval > 450 ms
* Receiving class Ia or class III antiarrhythmics

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Tisdale, PharmD, Principal Investigator — Purdue University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Tisdale JE, Wroblewski HA, Wall DS, Rieger KM, Hammoud ZT, Young JV, Kesler KA. A randomized, controlled study of amiodarone for prevention of atrial fibrillation after transthoracic esophagectomy. J Thorac Cardiovasc Surg. 2010 Jul;140(1):45-51. doi: 10.1016/j.jtcvs.2010.01.026. Epub 2010 Apr 9. PMID 20381077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2004 and November 2008, 80 patients were enrolled in the study, with 40 patients randomized to each arm. Patients were recruited from an academic medical center prior to undergoing esophageal surgery
Pre-assignment Details: 133 patients were screened for eligibility. 39 were excluded prior to consent d/t presence of exclusion criteria or declined participation. 94 were consented. 14 did not participate: 3 had pre-op exclusion criteria; 4 were withdrawn because the study protocol was delayed; 7 were excluded because they developed intra-operative atrial fibrillation
Groups:
- Control: Control usual care
Period: Overall Study
Arm/Group | Amiodarone | Control
Started | 40 | 40
Completed | 38 (40 completed analysis) | 40
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amiodarone | Control | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 43
  >=65 years | 18 | 19 | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (10) | 63 (9) | 62 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 34 | 33 | 67
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Atrial Fibrillation
Time Frame: 7 days
Population: Analysis was per protocol
Measure: Number; unit: participants
Arm/Group | Amiodarone | Control
Number analyzed (Participants) | 40 | 40
participants | 6 | 16
Statistical Analysis 1: Comparison: Amiodarone vs Control; Test type: Superiority or Other; p = 0.02, Chi-squared; Risk Ratio (RR) = 0.38, 95% CI 2-sided [0.16 to 0.86]

2. Secondary Outcome: Length of Post-surgical Hospital Stay
Time Frame: Duration of hospitalization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Amiodarone | Control
Number analyzed (Participants) | 40 | 40
days | 11 [9 to 15] | 12 [9.5 to 15]
Statistical Analysis 1: Comparison: Amiodarone vs Control; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Length of Post-surgical Intensive Care Unit Stay
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Amiodarone | Control
Number analyzed (Participants) | 40 | 40
hours | 68 [38 to 124] | 77 [39 to 122]
Statistical Analysis 1: Comparison: Amiodarone vs Control; Test type: Superiority or Other; p = 0.097, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants With Adverse Effects
Description: Adverse effects, including cardiovascular (hypotension, bradycardia, prolonged QT interval, ventricular tachycardia), respiratory (ARDS, pneumonia, atelectasis), and other (pericardial effusions, anastomotic leak)
Time Frame: 7 days
Population: Per protocol
Measure: Number; unit: patients
Arm/Group | Amiodarone | Control
Number analyzed (Participants) | 40 | 40
patients | 21 | 19
Statistical Analysis 1: Comparison: Amiodarone vs Control; Test type: Superiority or Other; p = 0.66, Chi-squared

ADVERSE EVENTS:
Arm/Group | Amiodarone | Control
Serious Adverse Events (participants affected / at risk) | 0/40 | 2/40
Other Adverse Events (participants affected / at risk) | 3/40 | 1/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amiodarone (N=40) | Control (N=40)
death (General disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amiodarone (N=40) | Control (N=40)
bradycardia (Cardiac disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Design not double-blind placebo-control Atrial fibrillation was left to discretion of treating MD Larger study necessary to determine differences in length of hospital stay and cost and identify infrequently occurring amiodarone adverse effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No